CLINICAL TRIAL: NCT03991884
Title: A Phase I Study of Dose-Adjusted Etoposide, Prednisone, Vincristine, Cyclophosphamide, and Doxorubicin Plus Escalating Doses of Inotuzumab Ozogamicin (DA-EPOCH-InO) in Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia
Brief Title: Inotuzumab Ozogamicin and Chemotherapy in Treating Patients With Recurrent or Refractory B-cell Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RG1004854; NCI-2019-03811 (Registry Identifier: NCI / CTRP); 8786 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Recurrent B Acute Lymphoblastic Leukemia; Recurrent B Lymphoblastic Lymphoma; Refractory B Acute Lymphoblastic Leukemia; Refractory B Lymphoblastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Etoposide; Doxorubicin; Vincristine; Prednisone; Cyclophosphamide; Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose -1 (0.3 mg/m^2) (Experimental): Patients receive etoposide, doxorubicin, and vincristine IV via continuous infusion on days 1-4, prednisone PO or IV BID on days 1-5, and cyclophosphamide IV over 1 hour on day 5. Patients also receive inotuzumab ozogamicin IV over 1 hour on day 8. Treatment repeats approximately every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Cyclophosphamide; Biological: Inotuzumab Ozogamicin
- Dose 1 (0.3 mg/m^2) (Experimental): Dose 1 patients receive etoposide, doxorubicin, and vincristine IV via continuous infusion on days 1-4, prednisone PO or IV BID on days 1-5, and cyclophosphamide IV over 1 hour on day 5. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 8 and 15. Treatment repeats approximately every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Cyclophosphamide; Biological: Inotuzumab Ozogamicin
- Dose 2 (0.6 mg/m^2, 0.3 mg/m^2) (Experimental): Dose 2 patients receive etoposide, doxorubicin, and vincristine IV via continuous infusion on days 1-4, prednisone PO or IV BID on days 1-5, and cyclophosphamide IV over 1 hour on day 5. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 8 and 15. Treatment repeats approximately every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Cyclophosphamide; Biological: Inotuzumab Ozogamicin
- Dose 3 (0.6 mg/m^2, 0.3 mg/m^2) (Experimental): Dose 3 patients receive etoposide, doxorubicin, and vincristine IV via continuous infusion on days 1-4, prednisone PO or IV BID on days 1-5, and cyclophosphamide IV over 1 hour on day 5. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 8 and 15. Treatment repeats approximately every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Cyclophosphamide; Biological: Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: Etoposide — Given IV
  Other Names: 33419-42-0; Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16; 141540
Drug: Doxorubicin — Given IV
  Other Names: 14-Hydroxydaunomycin; 23214-92-8; Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Vincristine — Given IV
  Other Names: 22-Oxovincaleukoblastine; LEUROCRISTINE; VCR; Vincrystine
Drug: Prednisone — Given PO or IV
  Other Names: 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Metacortandracin; Ofisolona; Orasone; Paracort; Predicor; Predicorten; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Cyclophosphamide — Given IV
  Other Names: Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclostin; Cyclostine; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: 635715-01-4; Besponsa; CMC-544; Way 207294; WAY-207294

SUMMARY:
This phase I trial studies the best dose of inotuzumab ozogamicin in combination with chemotherapy in treating patients with B-cell acute lymphoblastic leukemia that has come back (recurrent) or that does not respond to treatment (refractory). Inotuzumab ozogamicin is a monoclonal antibody, called inotuzumab, linked to a toxic agent called ozogamicin. Inotuzumab attaches to CD22 positive cancer cells in a targeted way and delivers ozogamicin to kill them. Drugs used in chemotherapy, such as etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving inotuzumab ozogamicin in combination with chemotherapy may kill more cancer cells than with chemotherapy alone in treating patients with recurrent or refractory B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
This is a dose-escalation study of inotuzumab ozogamicin.

Patients receive etoposide, doxorubicin, and vincristine intravenously (IV) via continuous infusion on days 1-4, prednisone orally (PO) or IV twice daily (BID) on days 1-5, and cyclophosphamide IV over 1 hour on day 5. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 8 and 15. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of CD22-positive, Philadelphia chromosome (Ph)-positive or Ph-negative B-cell acute lymphoblastic leukemia or lymphoblastic lymphoma. CD22 expression will be determined by multiparameter flow cytometry (MFC) or immunohistochemistry.
* Relapsed or refractory disease, as defined by any of the following:

  * Unable to achieve complete response (CR) despite >= 4 weeks of initial course of systemic therapy.
  * Recurrence of disease at any point after CR was achieved.

    * (Note: patients with Ph-positive disease must have received >= 1 second- or third-generation ABL kinase inhibitor as part of their prior treatment to be eligible.)
* Detectable disease, as defined by any of the following:

  * Presence of >= 5% abnormal blasts in the bone marrow or peripheral blood by morphology or MFC.
  * Patients with isolated extramedullary disease will be permitted if there is >= 1 site of disease that measures >= 1.5 cm in longest diameter on cross-sectional imaging.
* Absolute neutrophil count (ANC) >= 1,000/uL.
* Hemoglobin >= 8 g/dL.
* Platelets >= 50,000/uL.
* Note: Transfusions and growth factor support will be permitted within 3 days of initiation of study treatment to reach these thresholds. As patients with relapsed/refractory ALL frequently have cytopenias due to marrow infiltration by the disease, no hematologic parameters will be required for enrollment if cytopenias can be attributed to disease.
* Total serum bilirubin =< 1.5 x upper limit of normal (ULN); (unless due to Gilbert syndrome or hemolysis; =< 2 x ULN for hepatic abnormalities considered disease-related).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN.
* Serum creatinine =< 1.5 x ULN or serum creatinine level associated with a measured or calculated creatinine clearance of >= 40 mL/min.
* Corrected QT (QTc) interval =< 500 msec; if assessed, left ventricular ejection fraction >= 40%.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Must agree to the use of effective contraception while on study treatment, unless they are highly unlikely to conceive (defined as [1] surgically sterilized, or [2] women who are and men whose sexual partner[s] is/are postmenopausal [i.e., a woman who is > 50 years old or who has not had menses for >= 1 year], or [3] not heterosexually active for the duration of the study).

Exclusion Criteria:

* Patients with a circulating blast count of > 50,000/uL; systemic therapy with either hydroxyurea, vincristine, and/or corticosteroids will be permitted within 3 days of initiation of study treatment to reduce the blast count.
* Except for management of circulating blasts noted above, adequate duration from prior therapy must be achieved before initiation of study treatment, as defined below:

  * No cytotoxic or targeted systemic therapy < 2 weeks or 5 half-lives (whichever is shorter).
  * No blinatumomab < 2 weeks.
  * No radiation therapy < 4 weeks.
  * No monoclonal antibody therapy < 6 weeks (except for prior InO, as discussed below).
* Patients previously treated with InO will be eligible, unless they meet ANY of the following criteria:

  * > 6 individual doses (e.g., > 2 standard cycles) were administered.
  * Any documented hepatic toxicity observed was grade 3 or higher.
  * The most recent dose was administered < 3 months from the initiation of study treatment.
* For patients that have received prior allogeneic HCT, they must be >= 4 months from the date of stem cell infusion, with no prior history of sinusoidal obstruction syndrome/veno-occlusive disease (SOS/VOD), and off all treatment for graft-vs-host disease (GVHD) for >= 2 weeks. Patients with minimal active symptoms that can be controlled with topical therapies and/or the equivalent of prednisone =< 10 mg/day will be eligible.
* For patients that have received other forms of cellular immunotherapy (e.g., chimeric antigen receptor-modified [CAR] T cells), they must be >= 21 days from cell infusion, and any specific manifestations of cytokine release syndrome or neurologic toxicity attributable to the cellular therapy have completely resolved (i.e., < grade 1)
* Patients with a known history of chronic liver disease, including but not limited to cirrhosis, steatohepatitis, and chronic viral hepatitis. Patients with a history of GVHD of the liver will be permitted, provided they meet all of the other eligibility criteria.
* Patients with isolated testicular or central nervous system disease.
* Known hypersensitivity or intolerance to any of the agents under investigation.
* May not be pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of inotuzumab ozogamicin (InO) | Up to 5 years
  Will be defined as the highest dose of InO administered in which the incidence of dose limiting toxicities (DLTs) is < 33%, assuming at least 6 patients have been treated at this dose. DLTs assessed by:
  * Non-hematologic toxicities >= grade 3 evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 (except for febrile neutropenia/infection, unless felt to be a direct consequence of treatment-related toxicity [e.g., intestinal infection following mucosal barrier breakdown]).
  * Any instance of possible, probably, or definite SOS/VOD
  * Inability to complete 1 full cycle due to treatment-related adverse events
  * Any treatment delays > 3 weeks (i.e., to Day 50 of Cycle 1) for recovery of prolonged toxicity

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to 5 years
  Rate of complete response (CR) by bone marrow morphology and/or imaging.
Rate of complete minimal residual disease (MRD) response | Up to 5 years
  Assessed by multiparameter flow cytometry (MFC).
Progression-free survival | Up to 5 years
Relapse-free survival | Up to 5 years
Overall survival | Up to 5 years
Rate at which patients proceed to subsequent allogeneic hematopoietic cell transplantation (HCT) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Cassaday, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kopmar NE, Quach K, Gooley TA, Martino CH, Cherian S, Percival MM, Halpern AB, Ghiuzeli CM, Oehler VG, Abkowitz JL, Walter RB, Cassaday RD. Dose-Adjusted EPOCH Plus Inotuzumab Ozogamicin in Adults With Relapsed or Refractory B-Cell ALL: A Phase 1 Dose-Escalation Trial. JAMA Oncol. 2024 Jul 1;10(7):961-965. doi: 10.1001/jamaoncol.2024.0967. PMID 38722664

DOCUMENTS (1):
  • Informed Consent Form (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT03991884/ICF_000.pdf